CLINICAL TRIAL: NCT01058759
Title: Taxotere-Enoxaparin-(ENOXA)-Study: 1st-Line Docetaxel-Platin Chemotherapy as Single Therapy or in Combination With Enoxaparin in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer, a Phase III Study
Brief Title: Taxotere-Enoxaparin-(ENOXA)-Study
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The external funding (pharmaceutical company) was stopped and could not be substituded by internal funding.
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENOXA-NSCLC
Record Dates: First submitted 2010-01-28; First posted 2010-01-29 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: non-small cell lung cancer; NSCLC; Enoxaparin; Locally Advanced or Metastatic Non-small Cell Lung Cancer stadium IIIb/IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm B: Enoxaparin (Experimental)
  Interventions: Drug: Enoxaparin
- Arm A: No Enoxaparin (Active Comparator)
  Interventions: Other: No Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin
  Arms: Arm B: Enoxaparin
Other: No Enoxaparin
  Arms: Arm A: No Enoxaparin

SUMMARY:
Taxotere-Enoxaparin-(ENOXA)-Study: 1st-Line Docetaxel-Platin Chemotherapy as single therapy or in combination with Enoxaparin in patients aged older than 18 years with locally advanced or metastatic non-small cell lung cancer (stadium IIIb/IV), a phase III study. Study hypothesis: Increase of progressive free survival from 5 to 7.5 months.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Men and women aged 18 and older
* Locally Advanced or Metastatic Non-small Cell Lung Cancer stage IIIB/IV without any previous therapy
* Life expectancy at least 12 weeks
* EOCG performance < 1
* Appropriate renal and hepatic function
* Appropriate Hematology
* No bleeding events within 4 weeks prior to randomization
* No indication for prophylactic or therapeutic anticoagulation therapy
* Appropriate methods of contraception (both: men and women) for women of childbearing potential negative urine pregnancy test within 7 day prior to randomization
* Capability for s.c. injection of Enoxaparin every 24 hrs

Exclusion Criteria:

* History of cancer other than NSCLC
* Known contraindication for Enoxaparin e.g. HIT,
* Known contraindication for Docetaxel, Cisplatin, Carboplatin or co-medication
* Participation in any other clinical trials within 30 days prior to randomization
* Any known medical condition that does not allow therapy according to study protocol
* Seizure disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-11; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Progressive free survival | monthly

SECONDARY OUTCOMES:
Overall survival | monthly
RECIST | monthly
Quality of life | every three months
thromboembolic complications | monthly
safety of long term application of Enoxaparin | monthly
overall toxicity | monthly

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Dickgreber, MD, Study Chair — Hannover Medical School
Locations (1):
- Hannover Medical School, Department of Pneumology, Hanover, Lower Saxonia, Germany